CLINICAL TRIAL: NCT01407185
Title: Efficacy of a Home-Based Exercise Program in the Management of Heart Failure: An Evidenced-Based Multi-Disciplinary Approach
Brief Title: Efficacy of a Home-Based Exercise Program for Heart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment. Difficult to obtain Physician approval.
Sponsor: Catholic Home Care (Other)
Collaborators: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Kenneth L Miller, PT, DPT, Co-Principal Investigator, Catholic Home Care
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011_HF_STUDY
Record Dates: First submitted 2011-07-27; First posted 2011-08-02 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Heart Failure
Keywords: heart failure; quality of life; fall prevention; endurance; resistive training
MeSH Terms: conditions — Heart Failure | interventions — Exercise; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resistive Training (Experimental): Subjects will be working at 30-60% of 1 RM. The therapist selects theraband that will produce muscle fatigue ~ 15 reps. Subjects should report that the exercise was somewhat light to somewhat hard 11 to 14 on RPE scale. Increase or decrease resistance until the desired RPE is obtained. Continues until momentary fatigue is evidenced. Fatigue is defined as the inability to move through the full ROM in a slow controlled fashion. Record the exercise performed, amount of resistance, and # of good quality reps performed before fatigue was reached. A single set will be done for each muscle group.
  Interventions: Other: Resistive Exercise Training

INTERVENTIONS:
Other: Resistive Exercise Training — Resistive Exercises (between 8 and 12 exercises for both upper and lower body) at 30 to 60% of 1 RM for 2x per week for 12 months.
  Other Names: exercise training; physical therapy

SUMMARY:
The purpose of this study is to determine the efficacy of a multi-disciplinary home program consisting of specific education and home-based individualized combined aerobic and resistance training exercise program for persons with heart failure (NYHA class II-III). The investigators will assess effects on endurance, gait speed, lower extremity strength, hospital re-admission rate and the quality of life in community-dwelling older adults from 60 - 85 years of age over a 12 month period.

Anticipated Results: The researchers expect confirm their hypothesis that there will be a statistically significant difference between the experimental group receiving the combined aerobic and resistance training program and the control group receiving usual care based on strength, endurance, quality of life, falls, and hospital re-admission data.

DETAILED DESCRIPTION:
This study is IRB approved at Catholic Home Care and at New York Institute of Technology due to collaboration between Catholic Home Care and New York Institute of Technology. Subjects will be volunteers, recruited during the initial therapy visit from 10 trained CHC staff and subsequently randomized based on their patient identification number into an experimental group or experimental group after consent has been obtained.

Subjects will sign a consent form to enter the study. Two groups of 40 subjects will be required to finish in order to obtain power of 80 at an alpha of .05. The subjects will be living at home with a reliable caregiver. The nurse will provide current best practice to all CHF patients in the study which includes educating the patient and caregiver regarding diet, medication regime, monitoring for signs and symptoms to report and provide coordination of other disciplines such as social work for those with depression requiring additional management during OASIS screening.

During the initial physical therapy visit, the usual care assessment will be performed, in addition, to obtaining pre-test baseline data for the experimental and control groups. A preliminary home exercise program will be assigned. A handout on pacing activity and deep breathing will be given. The importance of and reason for the perceived exertion scale will be explained to experimental group subjects and a handout will be given that will be part of the study packet.

All subjects will be encouraged to complete the home aerobic portion a minimum of 2 times per day and will be given an activity log from which to check off the same and enter the number and distance achieved when walking for exercise. Resistance exercises will be done at least twice per week with one day of rest between sessions. For the control group subsequent sessions will include usual home care physical therapy consisting of breathing exercises, therapeutic exercise, transfer, gait training, and home exercise programs. Baseline measurements (field testing) will be completed at the initial evaluation and discharge from therapy. In addition, the Minnesota Living with Heart Failure Questionnaire (MLHFQ), and questions about re-hospitalizations, activity logs, falls follow up will be collected and reviewed at 6 and 12 months after the program.

Baseline measurements: The 2-Minute step test (2MST) is an aerobic measure that has been used with older adults.17 The subject is instructed to raise the knee joint to a point halfway between the patella and iliac crest at a comfortable pace for 2 minutes. It is scored by counting the number of times the right knee reaches the point described for 2 minutes. Vital signs including BP, PR, RR, RPE, pulse ox, and signs and symptoms of decompensation are monitored before, during and after test administration. The 2MST has been validated to several other measurement tools of aerobic capacity/endurance.

The MLHFQ is a self report outcome tool that measures the quality of life (QoL) in people with CHF. The MLHFQ is a widely used QoL assessment tool. Although the MLHFQ incorporates relevant aspects of three dimensions of quality of life, the questionnaire was not designed to measure any particular dimension separately. The total score should be taken as the best measure of how heart failure and treatments impact an individual's quality of life.21 The MLHFQ differentiated New York Heart Association Functional groups.

The 30 second chair rise test assesses lower extremity strength and endurance.20, 23,24 Jones et al report having a moderately high correlation between chair stand performance and maximum weight-adjusted leg press performance for both men and women (r=.78 and .71 respectively) supporting the criterion-related validity of the chair stand test as a measure of lower extremity strength.

Gait speed is a powerful tool that can have predictive value. Cesari et al reported that gait speed of less than 1 m/sec identifies persons at high risk of health-related outcomes including mortality and physical disability in well-functioning older people.26 Montero-Odasso et al found that gait speed is also predictive of adverse health-related outcomes in well-functioning elderly persons and recommend it be considered as a "vital sign".27 Hardy et al reported that improvements in gait speed predict a substantial reduction in mortality.28 Studenski et al reported that gait speed of less than .6 m/sec is predictive for future risk of hospitalization and decline in health and function.29 We will use comfortable gait speed. Normative data has been provided for both comfortable gait speed and fast gait speed by Bohannon and Lusardi et al..30, 31, 32, 33 For the experimental group, subsequent visits will include the monitoring of ital signs, activity log, progressing aerobic and resisted exercise using elastic tubing.

Aerobic exercise protocol (will be performed in subject's home):

The aerobic component of this study will be based on the tolerance of the subject and based on the vital signs, Pulse Oximetry, and RPE. These parameters will be reassessed after walking activity. Any subject that is not responding appropriately will not continue that day and a telephone call will be made to the MD following CHC's protocol for physician notification based on vital signs and signs and symptoms .

The subject will use assistive devices as necessary. During therapy sessions there will be a focus on pacing and improving any deviations noted. A distance baseline will determined the first visit. The home walking program will be done at least twice a day, preferably building up to an hourly frequency, with caregiver supervision or assist as necessary. The instructions for the patient will be to walk until slightly fatigued, preferably reaching an RPE of 11-14 and increasing their ambulation distance over time.

Resistance training protocol:

All subjects will be working at 30-60% of 1 RM. In general, therapists will provide the necessary guidance to insure that the postural base is sound, there is good stabilization, and no substitutions are occurring. All subjects will be monitored for vital signs before and after program and during program as needed, based on signs, symptoms and patient complaints for decompensation.

Intensity

1. The therapist selects theraband that will produce muscle fatigue ~ 15 repetitions.
2. Have the subject perform 1-2 repetitions. Moving at a slower speed will allow for greater control and less chance of injuries. Tell the patient that they should be able to stop on the dime when exercising.
3. The subject should report that the exercise was somewhat light to somewhat hard.
4. If the subject reports that it is less fairly light, increase resistance.
5. If the subject rates it as somewhat hard or more reduce the resistance.
6. Repeat until the desired RPE is obtained.
7. The exercise continues until momentary fatigue is evidenced. Fatigue is evidenced by noting an increased speed of movement to overcome resistance, followed by the inability to complete the repetitions when prompted to slow down. In this case the exercise is complete. Also fatigue is achieved when the exerciser is unable to complete reps when prompted to maintain good form.
8. Fatigue is therefore defined as the inability to move through the full ROM in a slow controlled fashion. Since you have achieved fatigue; 1 set is sufficient.
9. Record the exercise performed, amount of resistance, and # of good quality reps performed before fatigue was reached. A single set will be done for each muscle group14 Progression

1. If the subject was able to complete 25+ repetitions of an exercise the prior session for a given muscle group, increase the resistance 10% 2. If the subject completed < 25 reps keep the resistance the same 3. Repeat the same sequence for all subsequent sessions. Continue to document the amount of resistance used and the number of reps each exercise.

Duration: the duration for the therapist supervised portion of the program is shorter than comparable studies in the literature. However, the frequency and duration match current practice patterns in home care.

1. Allow frequent rests.
2. Should not be longer than 30 minutes to start. Frequency: weeks 1 and 2 will have a frequency of: 2-3x/week each week and week 3 and all subsequent weeks will have a frequency of 2x/week. It is anticipated that almost all subjects will have achieved functional goals and finish their PT home care in 4 weeks. Subjects will continue at 2x per week upon discharge with their caregiver. The subject and caregiver will be trained in RPE and symptom monitoring for decompensation.
3. Moving slowly reduces the need for stretching.
4. Explain to the subject that physical activity may make them feel soreness or achiness, but this is a normal and expected response to exercise.
5. It is expected that the patients will be doing the resistance exercises twice each week with a rest day in between. Aerobic programming will be done at least 2 times each day building up to hourly with the walking program.

Follow up: All participants will receive a telephone call from a physical therapist that is blinded to group assignment at 6 and 12 months that will complete the MLHFQ, take a falls history, and ask about subsequent hospitalizations. Activity logs will be mailed in monthly. Participants will receive postage paid envelopes and receive phone calls as reminders monthly prior to required submission.

Statistics: All statistical analysis will be done using SPSS 15(SPSS Inc. Chicago, IL.). Differences between groups and changes over time baseline versus discharge will be assessed using a mixed design ANOVA. The independent variables are the interventions (experimental vs. control) and time is the repeated independent variable across all subjects. The dependent variables are: strength scores, 2-minute step test, Minnesota, Gait speed, chair stand test. Appropriate post hoc tests will be utilized in the event of significant finding in order to investigate pair wise effects. An alpha level of p<0.05 will be used for all statistical comparisons.

Research Design: This study will be a randomized, two group, experimental group (combined aerobic and resistance training) and control group (usual care), pre-post test design measuring the effects of a home-based combined aerobic and resistive training program with subjects between 60-85 years of age with chronic heart failure. The subjects will be evaluated at baseline and at 4 weeks for falls history, hospital re-admission history, endurance using the 2MST, quality of life using the MLHFQ, strength using the 30 second chair stand test, and comfortable gait speed for functional ability. The subjects will receive follow up phone call for falls, hospital re-admissions and MLHFQ at 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

On program at Catholic Home Care (CHC) Have a diagnosis of CHF NYHA II or III Medically stable 60 - 85 years of age at completion of study Able to follow commands Normal vision (with corrective lenses, if necessary) Willing to participate in a program for 1 year Have a reliable caregiver that is willing to assist as necessary -

Exclusion Criteria:Latex allergy, Unstable CHF NYHA IV Pain that interferes with activity Active neurological and or orthopedic problems, Cancer, End stage renal disease Decreased balance as indicated on Tinetti balance assessment < 10/16.

-

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life | There is expected to be a change along each time point from Baseline to 4 weeks, 6 months, 12 months
  Minnesota Living with Heart Failure Questionnaire

SECONDARY OUTCOMES:
Re-hospitalization rates | 6 months, 12 months
  Telephone survey for hospitalization incidence from discharge to 12 months.
Falls incidence | 6 Months, 12 Months
  Telephone survey of falls incidence from discharge to 12 months.
Aerobic Capacity/Endurance | Baseline, subjects will be followed through duration of intervention for an average of 4 weeks
  2 Minute Step Test
Lower Extremity Strength | Baseline, subjects will be followed through duration of intervention for an average of 4 weeks
  30 Second Chair Stand Test
Gait Speed | Baseline, subjects will be followed through duration of intervention for an average of 4 weeks
  Gait speed is a tool that has predictive value. Gait speed identifies persons at high risk of health-related outcomes including mortality and physical disability in well-functioning older people. Gait speed also predicts falls risk, future hospitalization risk and decline in health and status.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Miller, PT, DPT, Principal Investigator — Catholic Home Care; Veronica Southard, DHSc, Principal Investigator — New York Institute of Technology and Catholic Home Care
Locations (1):
- Catholic Home Care, Holtsville, New York, United States